CLINICAL TRIAL: NCT02872753
Title: Intra-operative ACP Injection Following Partial Meniscectomy: a Randomized Controlled Trial
Brief Title: Intra-operative Injection of Autologous Conditioned Plasma (ACP) Following Partial Meniscectomy
Acronym: ACP-MEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACP-MEN
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2022-09

CONDITIONS: Meniscectomy
Keywords: Autologous Conditioned Plasma; meniscectomy; randomized controlled trial; intra-op injection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACP GROUP (Experimental): Patients will receive a single intra-op ACP injection following a procedure of arthroscopic partial meniscectomy (medial or lateral)
  Interventions: Biological: ACP
- CONTROL GROUP (Other): Patients will be treated by standard meniscectomy alone (medial or lateral)
  Interventions: Other: Standard Meniscectomy

INTERVENTIONS:
Biological: ACP — Autologous Conditioned Plasma will be obtained directly in the operatory room from the peripheral venous blood of the patient, and injected intra-articularly at the end of arthroscopic meniscectomy
  Arms: ACP GROUP
Other: Standard Meniscectomy — Patients will receive standard arthroscopic meniscectomy
  Arms: CONTROL GROUP

SUMMARY:
The aim of the present double blind controlled study is to evaluate the effects in terms of pain control and functional recovery provided by a single intra-operative injection of ACP performed at the end of arthroscopic partial meniscectomy.

Patients included in this trial will be randomized in two treatment groups: the first one will receive a single injection of 3-5 cc of ACP (using a dedicated centrifuge) at the end of the arthroscopic meniscectomy, whereas the second group will be treated by surgery alone. In order to ensure the double blinding of the trial all the patients enrolled will undergo blood harvesting before anesthesia, and acp will be produced just for the patients included in ACP group.

All patients will be evaluated basally, and then at 15, 30, 60, and 180 days after surgery by the following evaluation tools: IKDC (International Knee Documentation Committee) subjective, VAS (Visual Analogue Score) for pain, EQ-VAS for general Health Status, KOOS (Knee Injury and Osteoarthritis Outcome Score) and Tegner score. Furthermore, during the basal evaluation and at each follow-up visit up to 2 months, active and passive Range of Motion (ROM) of both the operated and contralateral knee were documented; also in addition, the trans-patellar circumference of both knees was registered to assess the trend of knee swelling over time.

Drugs assumption during the follow-up period will be recorded for each patient. All eventual adverse events occurred during the follow-up period will be registered.

ELIGIBILITY:
Inclusion Criteria:

* chronic symptomatic meniscal tears requiring partial resection;
* healthy contra-lateral knee (i.e. no pain or functional limitation in the contra-lateral joint);

Exclusion Criteria:

* meniscal lesions requiring suture;
* previous surgery on the index knee;
* other concurrent articular lesion requiring surgical treatment (e.g.: cartilage or ligament injuries);
* history of knee infectious arthritis;
* concurrent rheumatic, metabolic or severe systemic disease;
* Body Mass Index (BMI) > 30;
* known hypersensibility or allergy to/towards HA ;
* alcohol or other substances abuse/excess.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in IKDC (International Knee Documentation Committee) score over the various follow-up times | basal, 15,30,60,180 days
Change in VAS( Visual Analogue score) for pain over the various follow-up times | basal, 15,30,60,180 days

SECONDARY OUTCOMES:
Change in KOOS (Knee Injury and Osteoarthritis Outcome Score) over the various follow-up times | basal, 15,30,60,180 days
Change in Tegner Score over the various follow-up times | basal, 30,60,180 days
Change in transpatellar circumference over time | basal, 15,30,60,180 days
Change in active and passive ROM | basal, 15,30,60,180 days
Adverse events report | 15 days after surgery
Adverse events report | 30 days after surgery
Adverse events report | 60 days after surgery
Adverse events report | 180 days after surgery
Change in VAS for general health status | basal, 30,60,180 days

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Di Martino, MD, Study Director — Nano-biotechnology Lab, Rizzoli Orthopaedic Institute, Bologna, Italy; Giuseppe Filardo, MD, Principal Investigator — Biomechanics Lab, Rizzoli Orthopaedic Institute, Bologna, Italy; Berardo Di Matteo, MD, Study Chair — Biomechanics Lab, Rizzoli Orthopaedic Institute, Bologna, Italy
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams GD, Frank RM, Gupta AK, Harris JD, McCormick FM, Cole BJ. Trends in meniscus repair and meniscectomy in the United States, 2005-2011. Am J Sports Med. 2013 Oct;41(10):2333-9. doi: 10.1177/0363546513495641. Epub 2013 Jul 17. PMID 23863849
- [Background] Filardo G, Di Matteo B, Di Martino A, Merli ML, Cenacchi A, Fornasari P, Marcacci M, Kon E. Platelet-Rich Plasma Intra-articular Knee Injections Show No Superiority Versus Viscosupplementation: A Randomized Controlled Trial. Am J Sports Med. 2015 Jul;43(7):1575-82. doi: 10.1177/0363546515582027. Epub 2015 May 7. PMID 25952818
- [Background] Heard BJ, Barton KI, Chung M, Achari Y, Shrive NG, Frank CB, Hart DA. Single intra-articular dexamethasone injection immediately post-surgery in a rabbit model mitigates early inflammatory responses and post-traumatic osteoarthritis-like alterations. J Orthop Res. 2015 Dec;33(12):1826-34. doi: 10.1002/jor.22972. Epub 2015 Jul 7. PMID 26135713
- [Background] Thein R, Haviv B, Kidron A, Bronak S. Intra-articular injection of hyaluronic acid following arthroscopic partial meniscectomy of the knee. Orthopedics. 2010 Oct 11;33(10):724. doi: 10.3928/01477447-20100826-11. PMID 20954664
- [Background] Filardo G, Kon E, Roffi A, Di Matteo B, Merli ML, Marcacci M. Platelet-rich plasma: why intra-articular? A systematic review of preclinical studies and clinical evidence on PRP for joint degeneration. Knee Surg Sports Traumatol Arthrosc. 2015 Sep;23(9):2459-74. doi: 10.1007/s00167-013-2743-1. Epub 2013 Nov 26. PMID 24275957
- [Background] Andia I, Maffulli N. Platelet-rich plasma for managing pain and inflammation in osteoarthritis. Nat Rev Rheumatol. 2013 Dec;9(12):721-30. doi: 10.1038/nrrheum.2013.141. Epub 2013 Oct 1. PMID 24080861
- [Background] Boswell SG, Cole BJ, Sundman EA, Karas V, Fortier LA. Platelet-rich plasma: a milieu of bioactive factors. Arthroscopy. 2012 Mar;28(3):429-39. doi: 10.1016/j.arthro.2011.10.018. Epub 2012 Jan 28. PMID 22284405
- [Background] Lee HR, Shon OJ, Park SI, Kim HJ, Kim S, Ahn MW, Do SH. Platelet-Rich Plasma Increases the Levels of Catabolic Molecules and Cellular Dedifferentiation in the Meniscus of a Rabbit Model. Int J Mol Sci. 2016 Jan 16;17(1):120. doi: 10.3390/ijms17010120. PMID 26784189
- [Background] Blanke F, Vavken P, Haenle M, von Wehren L, Pagenstert G, Majewski M. Percutaneous injections of Platelet rich plasma for treatment of intrasubstance meniscal lesions. Muscles Ligaments Tendons J. 2015 Oct 20;5(3):162-6. doi: 10.11138/mltj/2015.5.3.162. eCollection 2015 Jul-Sep. PMID 26605189
- [Background] Pujol N, Salle De Chou E, Boisrenoult P, Beaufils P. Platelet-rich plasma for open meniscal repair in young patients: any benefit? Knee Surg Sports Traumatol Arthrosc. 2015 Jan;23(1):51-8. doi: 10.1007/s00167-014-3417-3. Epub 2014 Nov 7. PMID 25377191
- [Background] Griffin JW, Hadeed MM, Werner BC, Diduch DR, Carson EW, Miller MD. Platelet-rich plasma in meniscal repair: does augmentation improve surgical outcomes? Clin Orthop Relat Res. 2015 May;473(5):1665-72. doi: 10.1007/s11999-015-4170-8. Epub 2015 Feb 6. PMID 25663423
- [Derived] Lo Presti M, Costa GG, Agro G, Vasco C, Boffa A, Di Martino A, Andriolo L, Cenacchi A, Zaffagnini S, Filardo G. Platelet-Rich Plasma Injections Do Not Improve the Recovery After Arthroscopic Partial Meniscectomy: A Double-Blind Randomized Controlled Trial. Am J Sports Med. 2024 Nov;52(13):3198-3205. doi: 10.1177/03635465241283052. Epub 2024 Oct 18. PMID 39425245